CLINICAL TRIAL: NCT06093672
Title: Randomized, Open-label, Multicenter Phase 3 Study to Assess the Efficacy and Safety of GIVinostat Versus Hydroxyurea IN JAK2V617F-positive High-risk Polycythemia Vera Patients: the GIV-IN PV TRIAL
Brief Title: Study on Efficacy and Safety of Givinostat Versus Hydroxyurea in Patients With Polycythemia Vera
Acronym: GIV-IN-PV
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Italfarmaco (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DSC/08/2357/32; 2022-502276-23-00 (EU CTIS Number)
Record Dates: First submitted 2023-10-10; First posted 2023-10-23 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Polycythemia Vera
Keywords: Polycythemia Vera; Givinostat
MeSH Terms: conditions — Polycythemia Vera | interventions — givinostat; givinostat hydrochloride; Hydroxyurea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Givinostat - Core phase (Experimental): Givinostat 50 mg BID from baseline till week 48
  Interventions: Drug: Givinostat
- Hydroxyurea - Core phase (Active Comparator): HU 500 mg BID from baseline till week 48
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Givinostat — Oral. The dosage must be modified, according to the manifestation of toxicities or lack of efficacy, with the aim to achieve an optimized dose.
  Other Names: ITF2357
  Arms: Givinostat - Core phase
Drug: Hydroxyurea — Oral. The dosage must be modified, according to the manifestation of toxicities or lack of efficacy, with the aim to achieve an optimized dose.
  Other Names: ITF2357
  Arms: Hydroxyurea - Core phase

SUMMARY:
The goal of this clinical trial is to compare the efficacy and safety of givinostat to hydroxyurea in Jak2V617F-positive high risk polycythemia vera patients.

DETAILED DESCRIPTION:
PV is a cMPN mainly driven by JAK2V617F mutation. The disease has an increased risk of thromboembolic complications, a predisposition to evolve into myelofibrosis (MF) and transformation into acute myeloid leukemia.

Patients ≥ 60 years of age and/or with a previous thrombotic event (TE) are considered at High Risk (HR) for thrombosis. The association of absolute values of circulating neutrophil, lymphocyte and monocyte and the high value of JAK2V617F allele burden are additional risk factors for the occurrence of thrombosis and for progression to MF, respectively.

Overall, most patients treated with HU are not adequately under control for both symptoms and long-term risks.

In recent years, data have shown that histone deacetylase (HDACs) inhibitors induce growth arrest, differentiation, and/or apoptosis in neoplastic cells. Givinostat has demonstrated preliminary signs of clinical activity and an acceptable safety profile in patients with JAK2V617F-positive cMPNs in three phase 2 studies.

The core treatment phase (pivotal phase 3 study) is designed to demonstrate the superiority of givinostat versus HU on efficacy, in JAK2V617F-positive, HR PV patients.

The extended treatment phase will allow eligible patients to receive givinostat in the long-term, with the objective of collecting long-term safety and efficacy data.

ELIGIBILITY:
Core Treatment - Inclusion Criteria:

* Patients must have been diagnosed with PV according to the 2016 WHO criteria before randomization
* Patients must have JAK2V617F-positive disease
* Patients with PV must meet the definition of HR for thrombosis (i.e., HR) within 3 years before screening as follows:

  * Age ≥ 60 years, and/or
  * Prior thrombosis.
* Patients must be in need of treatment at screening, defined by the presence of at least one of the following:

  * HCT ≥ 45% or HCT < 45% with at least 1 phlebotomy performed in the 3 months before screening, or
  * WBC count > 10 × 109/L, or
  * PLT count > 400 × 109/L.
* Patients must have normalized HCT (i.e., HCT < 45%) at randomization

Extended Treatment - Inclusion Criteria

* Patients must have completed the Week 48 visit of the DSC/08/2357/32 core treatment phase and:

  1. if the patient received givinostat, a complete hematological response (CHR) at Week 48 shall be achieved
  2. if the patient received HU, did not achieve a CHR (see above for the definition) at Week 48

     Core Treatment phase - Exclusion Criteria
* Patients pre-treated with HU with a documented history of resistance or intolerance to HU defined by the original ELN criteria
* Patients with a QTcF value of > 450 msec for males and > 460 msec for females at the Screening visit (as the mean of 3 consecutive readings 5 minutes apart in the event a first ECG demonstrates a prolonged QTcF interval); congenital or acquired history of QTc prolongation or ventricular arrhythmias, at the Screening visit
* Splanchnic thrombosis and/or thrombosis of the cerebral venous sinuses and/or splenectomy in the medical history
* Patients with clinically significant cardiovascular disease
* Patients with myocardial infarction, stroke or unstable angina within the 6 months prior to screening.
* Patients with inadequate liver or renal function at screening
* Uncontrolled hypertriglyceridemia at screening, i.e., triglycerides ˃ 1.5 × ULN
* Previous treatment with a JAK2 or HDAC inhibitor or 32-phosphorus (radioactive isotope) therapy.
* Patients being treated concurrently with any investigational agent or prior participation in an interventional clinical study within the 30 days prior to screening or within 5 half-lives of the investigational product, whichever is longer.
* Pregnant or nursing women

Extended treatment phase - Exclusion criteria

* For patients randomized to givinostat in the core treatment phase - Patients with a QTcF value at Week 48 of > 500 msec
* For patients randomized to HU in the core treatment phase:

  * PLT count ≤ 150 × 109/L at Week 48
  * ANC < 1.2 × 109/L at Week 48
  * Uncontrolled hypertriglyceridemia at Week 48
  * Patients with a QTcF value at Week 48 of > 450 msec for males and > 460 msec for female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving a response at Week 48. | week 25 - week 48
  Response assessment based on:
  * Hematocrit < 45% without phlebotomy in the prior 3 months, and
  * White blood cell (WBC) count ≤ 10 × 109/L, and
  * Platelet count ≤ 400 × 109/L, and
  * Normal spleen size as measured by imaging (normal spleen size is defined as: a longitudinal diameter ≤ 12 cm for female and ≤ 13 cm for male) and
  * During Part 2 (Week 25 to 48), absence of progressive disease, major hemorrhagic events and major thrombotic events.

SECONDARY OUTCOMES:
Proportion of patients achieving a complete hematological response (CHR) at Week 48. | week 48
  CHR based on:
  * Hematocrit < 45% without phlebotomy in the prior 3 months, and
  * White blood cell (WBC) count ≤ 10 × 109/L, and
  * Platelet count ≤ 400 × 109/L
Time from randomization to the first observed CHR | Randomization - week 48
Proportion of patients with a normal spleen size at Week 48. | week 48
Safety and tolerability up to Week 48. | Randomization - week 48

CONTACTS AND LOCATIONS:
Locations (82):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Emad Ibrahim, MD, Inc, Redlands, California
  - US Oncology Inc, Englewood, Colorado
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Oncology Associates of Oregon, P.C., Eugene, Oregon
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology (Webster) - USOR, Houston, Texas
  - Texas Oncology-Denison Cancer Center, Sherman, Texas
  - University of Utah - Huntsman Cancer Institute - PPDS, Salt Lake City, Utah
  - The James Cancer Hospital and Solove Research Institute, Roanoke, Virginia
  - VA Puget Sound Health Care System - NAVREF - PPDS, Seattle, Washington
- Austria (4):
  - Landesklinikum Wiener Neustadt, Wiener Neustadt, Lower Austria
  - Ordensklinikum Linz GmbH Elisabethinen, Linz, Upper Austria
  - Klinikum Wels-Grieskirchen GmbH, Wels, Upper Austria
  - Medizinische Universitat Wien (Medical University of Vienna), Vienna, Vienna
- Bulgaria (3):
  - Acibadem City Clinic Multiprofile Hospital for Active Treatment Tokuda, Sofia, Sofia-Grad
  - University Multiprofile Hospital for Active Treatment Sveti Georgi EAD, Plovdiv
  - University Multiprofile Hospital for Active Treatment - Prof. Dr. Stoyan Kirkovich AD, Stara Zagora
- Croatia (4):
  - Clinical Hospital Dubrava, Zagreb, City of Zagreb
  - Clinical Hospital Center Rijeka - PPDS, Rijeka
  - Clinical Hospital Center Rijeka, Rijeka
  - General Hospital Sibenik, Šibenik
- France (9):
  - Centre Hospitalier de Saint-Quentin, Saint-Quentin, Aisne
  - CHU de Nice, Nice, Alpes-Maritimes
  - Centre Hospitalier de Troyes, Troyes, Aube
  - Hôpital Bretonneau, Tours, Indre-et-Loire
  - CHU Nantes, Nantes, Loire-Atlantique
  - CHU Angers, Angers, Maine-et-Loire
  - CHU Amiens Hôpital Sud, Amiens, Somme
  - Hôpital Saint Louis, Paris
  - Hopital d'Argenteuil, Argenteuil, Île-de-France Region
- Germany (4):
  - Medizinische Fakultät Mannheim der Universität Heidelberg, Universitätsmedizin Mannheim, Mannheim, Baden-Wurttemberg
  - Gemeinschaftspraxis Hämatologie - Onkologie, Dresden, Saxony
  - Universitätsmedizin Halle, Universitätsklinikum Halle, Klinik für Innere Medizin IV, Halle, Saxony-Anhalt
  - OncoResearch Lerchenfeld GmbH, Hamburg
- Hungary (3):
  - Gyor-Moson-Sopron Vármegyei Petz Aladár Egyetemi Oktató Kórház, Győr, Győr-Moson-Sopron
  - Szabolcs-Szatmár-Bereg Vármegyei Oktatókórház, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Tolna Vármegyei Megyei Balassa János Kórház, Szekszárd, Tolna County
- Ireland (3):
  - Cork University Hospital, Cork
  - Connolly Hospital Blanchardstown, Dublin
  - Mater Misericordiae University Hospital, Dublin
- Israel (4):
  - Hadassah Medical Center - PPDS, Jerusalem, Jerusalem
  - Assuta Medical Center, Tel Aviv, Tel Aviv
  - Bnai Zion Medical Center, Haifa
  - Carmel Medical Center, Haifa
- Italy (16):
  - Istituto Tumori "Giovanni Paolo II" I.R.C.C.S., Bari, Apulia
  - Grande Ospedale Metropolitano Bianchi-Melacrino-Morelli, Reggio Calabria, Calabria
  - Azienda Ospedaliero-Universitaria Di Bologna IRCCS Istituto Di Ricerca E Di Cura A Carattere Scientifico, Bologna, Emilia-Romagna
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST S.r.l, Meldola, Emilia-Romagna
  - Azienda USL IRCCS di Reggio Emilia, Reggio Emilia, Emilia-Romagna
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine, Friuli Venezia Giulia
  - Fondazione Policlinico Universitario Campus Bio-Medico di Roma, Rome, Lazio
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo, Lombardy
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Azienda Sanitaria Ospedaliera S. Croce e Carle, Cuneo, Piedmont
  - A.O.U. Maggiore della Carità, Novara, Piedmont
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Turin, Piedmont
  - Azienda Ospedaliero Universitaria Policlinico G Rodolico San Marco di Catania, Catania, Sicily
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo, Sicily
  - Azienda Ospedaliero Universitaria delle Marche, Ancona, The Marches
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
- Netherlands (3):
  - Spaarne Gasthuis, Hoofddorp, North Holland
  - Medisch Spectrum Twente, Enschede, Overijssel
  - Albert Schweitzer Ziekenhuis, Dordrecht, South Holland
- Poland (3):
  - Indywidualna Specjalistyczna Praktyka Lekarska Tomasz Woźny, Poznan
  - Specjalistyczny Szpital im. dra Alfreda Sokołowskiego, Wałbrzych
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza- Radeckiego we Wrocławiu, Wroclaw
- Serbia (5):
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Clinical Hospital Center Zemun, Belgrade
  - University Clinical Center of Serbia, Belgrade
  - University Clinical Center Nis, Niš
  - Clinical Center of Vojvodina, Novi Sad
- Spain (5):
  - ICO Badalona-H.U. Germans Trias i Pujol, Badalona, Barcelona
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- United Kingdom (2):
  - Belfast City Hospital, Belfast
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: No